CLINICAL TRIAL: NCT00571831
Title: The Effect of a Blue Light Filtering Intraocular Lens on Blood Retinal Barrier After Cataract Surgery
Brief Title: The Effect of a Blue Light Filtering IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa University (Other)
Responsible Party: Toshihiko Ueda/Associate Professor, Dept. of Ophthalmology, School of Medicine, Showa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Toshi-1; showa-IRB-02503
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: to Compare the Effect of Two Types of IOLs; on the Incidence of Cystoid Macular Edema; After Cataract Surgery
Keywords: macula edema; intraocular lens; prospective randomized parallel clinical design
MeSH Terms: interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- letter (No Intervention): a blue-filtering IOL an UV-filtering IOL
  Interventions: Procedure: intraocular lens implantation

INTERVENTIONS:
Procedure: intraocular lens implantation — Intraocular lens implantation
  Other Names: a blue-filtering IOL (ENV-13, Menicon Co.Ltd, Japan); an UV-filtering IOL (ES-13, Menicon Co.Ltd, Japan)

SUMMARY:
To compare the effect on blood retinal barrier disruption 3 and 12 months after implantation of either a blue light filtering intraocular lens(blue-filtering IOL) or an ultraviolet light filtering intraocular lens(UV-filtering IOL).

DETAILED DESCRIPTION:
The following parameters were measured for evaluation of blood retinal barrier disruption.

* the incidence of macular leakage by fluorescence angiography (FA)
* the mean fluorescein concentration in the vitreous by fluorophotometry (VFP)
* the thickness of the macula by optical coherence tomography (OCT)

Results

* the incidence fo macular leakage decreased significantly from 24%(3 months) to 5% (12 months) in the blue-filtering IOL group (P<0.05), and was significantly lower compared with the UV-filtering IOL group at 12 months.
* the VFP significantly decreased in both group from 3 to 12 months.
* the OCT decreased from 175 (3 months) to 166 um (12 months) in the blue- filtering IOL group.

ELIGIBILITY:
Inclusion Criteria:

* cataract patients
* All eligible for intraocular lens implantation

Exclusion Criteria:

* Patients had undergone an intraocular operation
* Patients had hypertensive retinopathy
* Patients had diabetic retinopathy
* Patients had ange-related macular degeneration
* no observable fundus
* The cataract operation was more than 30 minutes in duration

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-02; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To measure FA, VEP and OCT. | At 3 and 12 months after IOL implantation

CONTACTS AND LOCATIONS:
Overall Officials: Ryohei Koide, MD, PhD, Study Director — Department of Ophthalmology, School of Medicine, Showa University
Locations (1):
- Showa University Hospital, Tokyo, Tokyo, Japan